CLINICAL TRIAL: NCT05107050
Title: A Randomized Double-blind Controlled Clinical Trial Comparing a Synergistic Antimicrobial Cleanser and Gel to Normal Saline and an Amorphous Gel in Reducing Bioburden and Promoting Healing in Chronic Lower Extremity Ulcers
Brief Title: Comparing a Synergistic Antimicrobial Cleanser and Gel to Normal Saline and an Amorphous Gel in Reducing Bioburden and Promoting Healing in Chronic Lower Extremity Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Sanara MedTech (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIAKŌS
Record Dates: First submitted 2021-10-27; First posted 2021-11-04 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Wound of Skin

STUDY DESIGN:
Intervention Model Description: Randomized double-blind controlled clinical trial comparing a synergistic antimicrobial cleanser and gel to normal saline comparing to an amorphous gel in reducing bioburden and promoting healing in chronic lower extremity ulcers
Who Masked: Participant, Investigator
Masking Description: This protocol is double-blinded. Subjects will be randomized 1:1 to have their wound cleansed with either NSS-HG and AMC-AMG. Unblinded staff will prepare the solutions for the two arms the morning of the day of enrollment. NSS-HG and AMC-AMG will be placed in labeled containers consistent with the randomization scheme. Finally, the unblinded research staff will provide the subject with their 4-week supply of NSS-HG and AMC-AMG to take home. The unblinded staff will not assess the study ulcer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal saline wash and an amorphous gel (NSS-HG) (Active Comparator): Normal Saline Wash and Amorphous Gel
  Interventions: Device: Normal Saline and Amorphous gel
- synergistic antimicrobial cleanser (AMC) and antimicrobial gel (AMG) (Experimental): Antimicrobial Skin & Wound Cleanser helps in the mechanical removal of debris and foreign material from the skin, wound, or application site. BIAKOS™
  BIAKŌS Antimicrobial Wound Gel provides a moist environment to wound surfaces. BIAKŌS Antimicrobial Wound Gel is a safe and gentle colorless gel.
  Interventions: Device: BIAKOS™ Antimicrobial Skin & Wound Cleanser, BIAKŌS Antimicrobial Wound Gel

INTERVENTIONS:
Device: Normal Saline and Amorphous gel — Saline - sodium chloride and water Amorphous hydrogel dressings are formulations of water, polymers
  Arms: Normal saline wash and an amorphous gel (NSS-HG)
Device: BIAKOS™ Antimicrobial Skin & Wound Cleanser, BIAKŌS Antimicrobial Wound Gel — Antimicrobial Skin & Wound Cleanser helps in the mechanical removal of debris and foreign material from the skin, wound, or application site.
  BIAKŌS Antimicrobial Wound Gel provides a moist environment to wound surfaces. BIAKŌS Antimicrobial Wound Gel is a safe and gentle colorless gel. The gel provides preservative properties through the antimicrobial PHMB. BIAKŌS Antimicrobial Wound Gel: • Resists microbial colonization within the gel during shelf storage. • Provides an amorphous gel covering. • Facilitates autolytic debridement through a moist wound environment. Wounds experience some level of autolytic debridement in which the body's own enzymes breakdown necrotic tissue.
  Arms: synergistic antimicrobial cleanser (AMC) and antimicrobial gel (AMG)

SUMMARY:
The study is a randomized double-blind controlled clinical trial designed to compare healing rates between normal saline wash in combination with an amorphous gel (NSS-HG) versus the grouping of a synergistic antimicrobial cleanser (AMC) and antimicrobial gel (AMG) in chronic lower extremity ulcers.

After consenting, the ulcers of eligible subjects are measured, photographed and undergo the MolecuLight imaging procedure (MiX). The subject is then randomized to one of two arms: target ulcer cleansed saline wash and an amorphous gel (NSS-HG) or synergistic antimicrobial cleanser (AMC) and antimicrobial gel (AMG). After cleansing the wound a second MiX is performed. The subject is given a four-week supply.

DETAILED DESCRIPTION:
BIAKOS™ Antimicrobial Skin & Wound Cleanser helps in the mechanical removal of debris and foreign material from the skin, wound, or application site. BIAKOS™ Antimicrobial Skin and Wound Cleanser is a pure, colorless, isotonic cleanser that is safe. The preservative, PHMB, at a concentration of 0.1% w/w is added to the product to inhibit the growth of microorganisms such as Staphylococcus aureus, Staphylococcus epidermidis, Pseudomonas aeruginosa, Escherichia coli, antibiotic resistant Methicillin Resistant Staphylococcus aureus [MRSA). and fungus Candida albicans within the product.

BIAKŌS Antimicrobial Wound Gel provides a moist environment to wound surfaces. BIAKŌS Antimicrobial Wound Gel is a safe and gentle colorless gel. The gel provides preservative properties through the antimicrobial PHMB. BIAKŌS Antimicrobial Wound Gel: • Resists microbial colonization within the gel during shelf storage. • Provides an amorphous gel covering. • Facilitates autolytic debridement through a moist wound environment. Wounds experience some level of autolytic debridement in which the body's own enzymes breakdown necrotic tissue.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Presence of a diabetic foot ulcer, Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the tendon or muscle provided it is below the medial aspect of the malleolus OR Presence of a full thickness venous leg ulcer (VLU)
3. Index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to the initial screening visit.
4. Study ulcer size is a minimum of 0.75 cm2 and a maximum of 5 cm2 at first treatment visit for DFU OR a minimum of 2.0cm2 and a maximum of 20.0 cm2 at the first treatment visit for VLU.
5. Adequate circulation to the affected extremity as demonstrated by a transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, OR an Ankle Brachial Index (ABI - measure of blood flow to the ankle) between 0.7 and ≤ 1.3 OR a toe brachial index >0.5 within 3 months of the first Screening Visit.
6. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
7. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
8. Subject has read and signed the IRB approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

1. Study ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes or venous disease.
2. A surgery for operative debridement or revascularization is planned for the ulcer to be treated.
3. Index ulcer has a history of cancer or, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
4. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
5. History of radiation at the ulcer site.
6. Subject with DFUs who cannot adhere to strict offloading according to protocol standards in the opinion of the investigator.
7. Subjects with VLUs who cannot adhere to multilayer compression.
8. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
9. Active treatment of infection anywhere in the body with IV antibiotics, at screening and baseline.
10. Suspected or confirmed signs/symptoms of gangrene on any part of the affected limb.
11. Known Osteomyelitis or bone infection of the affected foot or leg as verified by diagnostic imaging within 30 days prior to enrollment.
12. Subject is pregnant or breast feeding.
13. Study ulcer with a history of treatment with hyperbaric oxygen, growth factors or other biologic treatments, or a Cellular or Tissue-based Product (CTP) within 30 days of enrollment.
14. Subject has a known or suspected allergy to products under study.
15. Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-25 (Estimated)

PRIMARY OUTCOMES:
Compare healing rates (percent area reduction) through digital device | 4-weeks
  Compare healing rates (percent area reduction) between normal saline wash and an amorphous gel (NSS-HG) to the combination of a synergistic antimicrobial cleanser (AMC) and antimicrobial gel (AMG) in chronic lower extremity ulcers.

SECONDARY OUTCOMES:
Compare the reduction in bacterial bioburden | 4-weeks
  Compare the reduction in bacterial bioburden as determined by the MolecuLight Procedure (MiX) between lower extremity ulcers treated with NSS-HG and AMC-AMG as determined by the WoundChek Protease Status between lower extremity ulcers treated with NSS-HG and AMC-AMG.
Pain Score | 4-weeks
  The difference in pain scores between subjects treated with NSS-HG and AMC-AMG using the numeric PEG score. The PEG scale is a validated pain scoring system. It consists of three 1-10 rating scales.
Adverse Events | 4-weeks
  Compare the difference in adverse events between subjects treated with NSS-HG and AMC-AMG determined by adverse event reporting through case report forms.

CONTACTS AND LOCATIONS:
Locations (1):
- The Serens Group Austin Research Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No